CLINICAL TRIAL: NCT05335200
Title: Radiation Dosimetry, Plasma Pharmacokinetics, Biodistribution, Safety and Diagnostic Performance of (S)-[18F]FBFP PET/CT in Healthy Volunteers and Patients With Central Nervous System Diseases
Brief Title: Clinical Applications of (S)-[18F]FBFP PET/CT in Healthy Volunteers and Patients With Central Nervous System Diseases
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM-SIGMA
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Patients With Central Nervous System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- (S)-[18F]FBFP injection and PET/CT scan (Experimental): Patients will be intravenously injected with(S)-[18F]FBFP and undergo PET/CT scan.
  Interventions: Diagnostic Test: (S)-[18F]FBFP PET/CT

INTERVENTIONS:
Diagnostic Test: (S)-[18F]FBFP PET/CT — Patients will be intravenously injected with 185-370MBq (S)-[18F]FBFP and undergo serial whole-body PET/CT scans at multiple time points (5min, 15min, 30min, 45min, 1h, 2h, 4h). Safety assessment and tolerability of the study will be conducted.

SUMMARY:
This is an open-label whole-body PET/CT (positron emission tomography/computed tomography) study for investigation of radiation dosimetry, plasma pharmacokinetics, biodistribution, safety and diagnostic performance of (S)-[18F]FBFP in healthy volunteers and patients with central nervous system diseases. A single dose of nearly 370 MBq (S)-[18F]FBFP will be intravenously injected into healthy volunteers and patients with central nervous system diseases. Visual and semiquantitative method will be used to assess the PET/CT images. Changes of blood pressure, pulse, respiration, temperature and any adverse events will be collected from the volunteers. Adverse events will also be observed in the patients.

DETAILED DESCRIPTION:
(S)-[18F]FBFP is a promising sigma-1 receptor radioligand. The sigma-1 receptor is a unique chaperone protein with 223 amino acids located at the mitochondria-associated endoplasmic reticulum membrane. Several lines of evidence have demonstrated that the sigma-1 receptor plays a pivotal role in the pathophysiology of many neuropsychiatric disorders including amyotrophic lateral sclerosis, Alzheimer's disease, Parkinson's disease, Huntington's disease, pain, depression and drug addiction.Therefore, it is an important target for the investigation of neuropsychiatric disorders and drug development. PET imaging of sigma-1 receptors in the human brain will enable the elucidation of this target's involvement in neurologic disorders and will also facilitate new drug development.

For further interests in clinical translation of PET sigma-1 receptors radioligands, (S)-[18F]FBFP, an open-label whole-body PET/CT study was designed to investigate radiation dosimetry, plasma pharmacokinetics, biodistribution, safety and diagnostic performance of (S)-[18F]FBFP in healthy volunteers and patients with central nervous system diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers: Males and females, ≥18 years old
* Patients With Central Nervous System Diseases: Patients with suspicion or diagnosis of central nervous system diseases after systemic neuropsychiatric assessment by experienced neurologists, having other imaging examination like CT or MRI, being able to provide basic information and sign the written informed consent form.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential
* Known severe allergy or hypersensitivity to [18F] radionuclides.
* Kidney or liver failure.
* Patients not able to enter the bore of the PET/CT scanner.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the Investigator, may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Visual and semiquantitative assessment of organs and biodistribution | 1 month
  Visual analysis will be performed by consensus reading by at least 3 experienced nuclear medicine physician. The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake values (SUVs) of lesions or organs will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, MD, Study Chair — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No